CLINICAL TRIAL: NCT06421571
Title: A Greek, Prospective Non-interventional Study Investigating the Effectiveness and the Mechanism of Action of Chlormethine (CL) Gel in the Treatment of MF-CTCL Adult Patients
Brief Title: The Mechanism of Action of Chlormethine (CL) Gel in the Treatment of MF-CTCL Adult Patients
Acronym: GR-CTCL_CL
Status: Recruiting | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: RECORDATI GROUP (Industry)
Responsible Party: Principal Investigator, Evangelia Papadavid, Professor, National and Kapodistrian University of Athens
Other Study IDs: 441/05-08-2020
Record Dates: First submitted 2024-03-26; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsies and blood from MF-CTCL patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chlormethine is a topical alkylating agent whose role in MF-CTCL has been extensively studied over the last 40 years. While its efficacy is well established, many safety concerns have been raised due to high rates of delayed cutaneous hypersensitivity to aqueous solutions that limit the prolonged use of chlormethine in clinical practice. It has been shown that complete response to topical chlormethine is associated with lower risk of disease progression. Accordingly, clinical data from the investigators' clinic confirm that chlormethine gel is a safe and effective treatment, which be used in early and advanced stages of cutaneous lymphomas. Based investigators' clinical and biological results , the investigators like to further investigate the change in the percentage as well as the profile of malignant and inflammatory cells by CyTOF analysis and further investigate the pathways (eg OX40, PDL1) involved in this process.

DETAILED DESCRIPTION:
1. RATIONALE Chlormethine is a topical alkylating agent whose role in MF-CTCL has been extensively studied over the last 40 years. While its efficacy is well established, many safety concerns have been raised due to high rates of delayed cutaneous hypersensitivity to aqueous solutions that limit the prolonged use of chlormethine in clinical practice. It has been shown that complete response to topical chlormethine is associated with lower risk of disease progression. Accordingly, the clinical data confirm that chlormethine gel is a safe and effective treatment, which be used in early and advanced stages of cutaneous lymphomas. In a study of 23 patients with stage IA-IIB mycosis fungoides from investigators' center an overall response of 65.22% at 9 months of treatment with topical chlormethine was recorded. Moreover in a recent multicenter greek study that included 58 patients with stage IA-IIB mycosis fungoides an overall response rate of 80.8% at 9 months of treatment was achieved. In the same study better response in patients with patches in comparison to plaques or tumors was also depicted. Unfortunately, the occurrence of skin drug reactions was the leading cause of treatment discontinuation in studies evaluating chlormethine irrespective of drug formulation, negatively affecting the achievement of a therapeutic response. In investigators' study, severe dermatitis was one of the main causes of treatment discontinuation, occuring in 15.5% of patients.

   Taper of application frequency (as per SmPC) and topical steroid use represent strategies allowing the management of dermatitis in order to maintain patients on CL gel treatment and prevent treatment discontinuation. The presence or severity of dermatitis in the study population was not associated with ORR, indicating that the development of dermatitis did not affect the likelihood of response. It has previously been suggested that dermatitis may be a prognostic indicator for clinical response. These data highlight the unmet need to explain the significance of dermatitis after topical chlomethine application and the immunological changes behind and how these affect the clinical response. Additionally by standardizing a CyTOF technique in CTCL samples from skin biopsies of CTCL patients, investigators established the methodology for identification and enumeration of different cells populations in situ and their interactions with tumor microenvironment. Investigators' preliminary data demonstrated that the evaluation of MF-CTCL patients' immune profile revealed differences in cell proportion pinpointing the heterogeneity that characterizes different stages of MF.

   Based on investigators' clinical and biological results investigators would like to further examine the change in the percentage as well as the profile of malignant and inflammatory cells by CyTOF analysis and further investigate the pathways (eg OX40, PDL1) involved in this process.
2. STUDY DESIGN 2.1 Study Description The proposed study is a non-interventional, prospective (data collection), open-label, single-arm study. Data collection will be done prospectively. The management of patients will be done in the classic framework of the management of adult patients with MF-CTCL in principal investigator's university hospital.
3. RESEARCH OBJECTIVES (CLINICAL, BIOLOGICAL AND PATIENT-REPORTED OUTCOMES - QUALITY OF LIFE) 3.1 Clinical objectives

   3.1.1 Effectiveness of CL gel treatment in routine medical practice in MF patients by:

   • Evaluation of clinical response by mSWAT
   * Duration of response (defined as the interval from the time measurement criteria for CR and PR are first met until the first date that progressive disease is documented), time to next treatment (TNTT: defined as the time from the time the next treatment is recorded)
   * Correlation between dermatitis occurrence and clinical response
   * quality of life of the patients
   * Chlormethine gel tube consumption
   * safety and tolerability of the treatment with CL gel: frequency of skin side effects 3.2 Biological objectives For this part of the study the percentage change of malignant and inflammatory cells, profile of inflammatory (new and existing) and malignant cells in all MF patients treated with chlormethine gel (with or without dermatitis), cytokines and signaling pathways at a single cell level will be also measured.

   3.2.1 Assessments Dermatitis occurrence (before any topical steroids application) Clinical response (at least score >50% improvement from baseline) At months 6 and 12
   * Evaluation of the impact of chlormethine gel treatment on malignant and inflammatory cells
   * Evaluation of the impact of chlormethine gel treatment exhibits on the profile of Th1/Th2 cytokines (ELISA)
   * Evaluation of the impact that CL gel treatment exerts on the JAK/STAT, NF-κB AKT, MAP signaling pathways (Western Blotting) 3.3 Patient-Reported Outcomes - quality of life (SKINDEX-29) Quality of Life (QoL) change from Baseline in the European Organization for Research and Treatment of Cancer (EORTC) Disease-Related Symptom Scales of the SKINDEX-29 at every visit.

   3.4 Study Population MF patients treated with CL gel as monotherapy. Study design is presented in figure below.

   This study will include 40 patients treated with CL gel as monotherapy.

   Patients will discontinue study treatment permanently if the following condition is met:

   • Patients are still unable to tolerate CL gel treatment at reduced frequency with co-administration of corticosteroids.

   All patients will be assessed every month for the first three months, and every 3 months thereafter (at months 6, 9, 12), as per current clinical practice.

   In case of dermatitis, the patient is encouraged to continue treatment with reduced frequency at every other day or every third day. Steroids will be used only if the reduced schedule is not sufficient. A temporary treatment interruption might occur for a period of 2 weeks and then treatment can be restarted.

   3.5 Research objectives (detailed) Clinical, biological and patient quality of life 3.5.1 Clinical objective

   • Effectiveness of CL gel treatment in routine medical practice in MF patients: Overall Response Rate (ORR), defined as the proportion of patients who achieved a CR or PR (at least score >50% improvement from baseline), in all patients determined by mSWAT, within 12 months of the start of CL gel treatment.
   * Duration of response (RD), time to next treatment (TNTT) in the framework of the trial
   * safety and tolerability of the drug: Frequency of skin side effects with a focus on dermatitis, the time to occurrence and duration of dermatitis as well as the percentage of patients with dermatitis remaining on treatment at the end of the study
   * Correlation between dermatitis occurrence and clinical response (ORR in patients experiencing or not dermatitis during treatment by chlormethine gel)
   * quality of life of the patients (using Skindex-29 tool) receiving CL gel for at baseline and at the end of treatment
   * Chlormethine gel tube consumption estimated from medical prescription and patients' statement 3.6 Biological objectives

   For this part of the study the percentage change of malignant and inflammatory cells, profile of inflammatory (new and existing) and malignant cells in all MF patients treated with chlormethine gel (with or without dermatitis), cytokines and signaling pathways at a single cell level will be also measured at:
   * Baseline

     o Dermatitis occurrence (before any topical steroids application)
     * Clinical response (at least score >50% improvement from baseline)
     * At months 6 and 12
   * Evaluation of the impact of chlormethine gel treatment on malignant and inflammatory cells using mass cytometry (CyTOF)
   * Evaluation of the impact of chlormethine gel treatment exhibits on the profile of Th1/ Th2 cytokines (ELISA)
   * Evaluation of the impact that CL gel treatment exerts on the JAK/STAT, NF-κB, AKT, MAP signalling pathways (western blot analysis)

   Skin histology description, immunohistochemistry and PCR are used in clinical routine practice to assess malignant T cells and clonality.

   The exploratory study will use both blood samples and skin biopsies taken as per routine management of the patients tests for the study of • CL gel mechanism of action (1)

   • the pathophysiology of dermatitis after CL gel application (2)

   We will correlate the above with the clinical effectiveness of CL gel treatment (3) as well as dermatitis occurrence and clinical response in MF patients (4).

   More specifically

   • the profile of malignant cells and inflammatory, by characterizing the immune cells deriving from single cell suspensions from biopsies and/or PBMCs by mass cytometry

   The signaling pathways involved, such as JAK/STAT, NF-κB, AKT, MAP kinases by identifying the phosphorylation status of implicated proteins by Western blot analyses

   3.7 Patient-Reported Outcomes - quality of life (SKINDEX-29) Definition: Quality of Life (QoL) change from Baseline in the European Organization for Research and Treatment of Cancer (EORTC) Disease-Related Symptom Scales of the SKINDEX-29 at every visit.

   The Skindex-29 is a skin disease-specific questionnaire that comprehensively assesses the effects of skin diseases on patient's quality of life. It was specifically developed to detect changes throughout time, as well as differences among patients with different skin diseases. The questionnaire covers areas considered crucial in an instrument designed to evaluate quality of life, such as: degree of symptoms, psychosocial functioning, and emotional status. The 29-item version is a refinement of a previous 61-item version. It was originally written in English and has already been translated and validated in other languages. The Skindex-29 inquiries about how often (Never, Rarely, Sometimes, Often, All the time) during the previous four weeks the patient experienced the effect described in each item. Seven items address the Symptoms domain, ten items the Emotional domain, and twelve items the Functioning domain. All responses are transformed to a linear scale of 100 varying from 0 (no effect) to 100 (effect experienced all the time). Skindex scores are reported as three scale scores, corresponding to the three domains; a scale score is the average of a patient's responses to items in a given domain.

   Five distinct categories for the Symptoms scale, and four for the Emotions and Functioning scales have been categorized as summarized in the table below:

   Emotional Symptoms Functioning Very little <6 <4 <4 Mild 6-24.9 4-10.9 4-10.9 Moderate 25-49.9 11-25.9 11-32.9 Severe ≥50 26-49.9 ≥33 Extreme ≥50

ELIGIBILITY:
Inclusion Criteria:

* MF-CTCL early-stage diagnosed patients, or late-stage patients that relapse without current active tumoral disease who still have patches and/or plaques.
* Age ≥ 18 years
* Patients naïve from CL gel treatment
* Early-stage patients who will be using CL as monotherapy: at enrolment without any concomitant MF treatment
* Early-stage patients if treated with other topical or systemic (late or early-stage patients) at enrolment, then a 2 week for topical steroids (and/or other topical treatment) and 4 weeks for systemic treatments wash out period will be required
* Women of child bearing potential must have a negative serum pregnancy test within 3 days prior enrolment.
* Women of child bearing potential should use adequate birth control measures, during the study treatment period until 30 days after treatment
* Women who are breast feeding should discontinue nursing prior to the first application of study treatment and until 30 days after the last study treatment
* Before patient enrolment, written informed consent must be given according to ICH/GCP

Exclusion Criteria:

* - Patients diagnosed with stage III and IV, unless they meet the inclusion criteria for late stage disease (see above)
* Patients with multiple active tumors - progressive disease
* Patients with concomitant and chronic use of topical or systemic corticosteroids for the treatment of any other disease
* Patients treated with concomitant topical (except chlormethine gel) and/or systemic MF treatments who have missed the wash-out period (2 weeks for topical treatment and 4 weeks for systemic treatment)
* Acute flare or atopic dermatitis or other dermatosis in the last 3 weeks
* Pregnant and breast-feeding women
* Patients unable to comply with study procedures (e.g. provide written consent, fill in the questionnaires, geographical condition potentially hampering compliance with the study protocol and follow-up schedule).
* Known hypersensitivity to any component of the CL gel formulation
* Concurrent or planned local or systemic anti-CTCL therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MF-CTCL patients, from outpatient PCL clinic from Attikon University Hospital, who will be candidates for topical treatment with chlormethine gel will be informed and invited to participate in this prospective data collection. All clinical and biological investigations (including blood samplings and biopsies) will be prescribed and arranged as part of standard routine clinical practice at PCL center.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical objectives: Number of participants with treatment-related adverse events as assessed by CTCAEv4.0. | 12 months
  Number of participants with treatment-related adverse events as assessed by CTCAEv4.0.
Clinical objectives: Clinical response mSWAT | 12 months
  Clinical response mSWAT (at least score ≥50% improvement from baseline) every month for the first three months, and every 3 months thereafter (at months 6, 9, 12), as per current clinical practice
Clinical objectives: Dermatitis occurrence | 12 months
  Dermatitis occurrence (before any topical steroids application)
Biological objectives: Evaluation of the impact of chlormethine gel treatment on malignant and inflammatory cells | 12 months
  Determine and compare immune cells vs malignant cells at single cell level
Biological objectives:Evaluation of the impact of chlormethine gel treatment exhibits on the profile of cytokines | 12 months
  Evaluation of the impact of chlormethine gel treatment exhibits on the profile of Th1/Th2 cytokines (ELISA)
Biological objectives:Evaluation of the impact that CL gel treatment exerts on the major signaling pathways | 12 months
  Evaluation of the impact that CL gel treatment exerts on the JAK/STAT, NF-κB AKT, MAP signaling pathways (Western Blotting)
Patient-Reported Outcomes | 12 months
  Questionnaires of Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- 1 Rimini Street, ATTIKON University Hospital, Athens, Greece

REFERENCES:
- [Result] Inturi S, Tewari-Singh N, Agarwal C, White CW, Agarwal R. Activation of DNA damage repair pathways in response to nitrogen mustard-induced DNA damage and toxicity in skin keratinocytes. Mutat Res. 2014 May-Jun;763-764:53-63. doi: 10.1016/j.mrfmmm.2014.04.002. Epub 2014 Apr 13. PMID 24732344
- [Result] Lessin SR, Duvic M, Guitart J, Pandya AG, Strober BE, Olsen EA, Hull CM, Knobler EH, Rook AH, Kim EJ, Naylor MF, Adelson DM, Kimball AB, Wood GS, Sundram U, Wu H, Kim YH. Topical chemotherapy in cutaneous T-cell lymphoma: positive results of a randomized, controlled, multicenter trial testing the efficacy and safety of a novel mechlorethamine, 0.02%, gel in mycosis fungoides. JAMA Dermatol. 2013 Jan;149(1):25-32. doi: 10.1001/2013.jamadermatol.541. PMID 23069814
- [Result] Kim EJ, Guitart J, Querfeld C, Girardi M, Musiek A, Akilov OE, Angello JT, Bailey WL, Geskin LJ. The PROVe Study: US Real-World Experience with Chlormethine/Mechlorethamine Gel in Combination with Other Therapies for Patients with Mycosis Fungoides Cutaneous T-Cell Lymphoma. Am J Clin Dermatol. 2021 May;22(3):407-414. doi: 10.1007/s40257-021-00591-x. Epub 2021 Mar 3. PMID 33656660
- [Result] Kim YH, Liu HL, Mraz-Gernhard S, Varghese A, Hoppe RT. Long-term outcome of 525 patients with mycosis fungoides and Sezary syndrome: clinical prognostic factors and risk for disease progression. Arch Dermatol. 2003 Jul;139(7):857-66. doi: 10.1001/archderm.139.7.857. PMID 12873880
- [Result] Kim YH, Martinez G, Varghese A, Hoppe RT. Topical nitrogen mustard in the management of mycosis fungoides: update of the Stanford experience. Arch Dermatol. 2003 Feb;139(2):165-73. doi: 10.1001/archderm.139.2.165. PMID 12588222
- [Result] Koumourtzis M, Lampadaki K, Dalamaga M, Papadavid E. Chlormethine Gel is Efficient and Safe in Mycosis Fungoides Skin Lesions. Acta Derm Venereol. 2022 Jun 9;102:adv00730. doi: 10.2340/actadv.v102.1095. PMID 35199177
- [Result] Lampadaki K, Koumourtzis M, Karagianni F, Marinos L, Papadavid E. Chlormethine Gel in Combination with Other Therapies in the Treatment of Patients with Mycosis Fungoides Cutaneous T Cell Lymphoma: Three Case Reports. Adv Ther. 2021 Jun;38(6):3455-3464. doi: 10.1007/s12325-021-01721-x. Epub 2021 Apr 30. PMID 33928511
- [Result] Papadavid E, Koumourtzis M, Nikolaou V, Lampadaki K, Marinos L, Patsatsi A, Georgiou E, Dalamaga M, Stratigos A. Chlormethine gel is effective for the treatment of skin lesions in patients with early- and late-stage mycosis fungoides in clinical practice. J Eur Acad Dermatol Venereol. 2022 Oct;36(10):1751-1757. doi: 10.1111/jdv.18183. Epub 2022 May 12. PMID 35470483
- [Result] Ramsay DL, Parnes RE, Dubin N. Response of mycosis fungoides to topical chemotherapy with mechlorethamine. Arch Dermatol. 1984 Dec;120(12):1585-90. PMID 6508330
- [Result] Querfeld C, Scarisbrick JJ, Assaf C, Guenova E, Bagot M, Ortiz-Romero PL, Quaglino P, Bonizzoni E, Hodak E. Post hoc Analysis of a Randomized, Controlled, Phase 2 Study to Assess Response Rates with Chlormethine/Mechlorethamine Gel in Patients with Stage IA-IIA Mycosis Fungoides. Dermatology. 2022;238(2):347-357. doi: 10.1159/000516138. Epub 2021 Jun 4. PMID 34091453
- [Result] Pavlidis A, Karagianni F, Vetsika EK, Koumourtzis M, Lampadaki K, Piperi C, Pappa V, Papadavid E. Bio-P-10 - Evaluation of the role of different cell populations in mycosis fungoides microenvironment as a tool for biomarker identification for disease progression and individualized therapy. EJC 2021:156(S1);S40-S41